CLINICAL TRIAL: NCT03162042
Title: Role of Myostatin, Activin A and Follistatin Cachexia of ENT Cancers
Acronym: MYOCACH
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-326; 2015-A00833-46 (Other: 2015-A00833-46)
Record Dates: First submitted 2017-05-05; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Cachexia; Squamous Cell Carcinoma; Head and Neck Cancer
Keywords: Activin A; Myostatin; Follistatin; Cachexia; Squamous cell carcinoma
MeSH Terms: conditions — Cachexia; Carcinoma, Squamous Cell; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Squamous cell carcinoma: 55 patients were included in the study : 32 in the cancer group (only squamous cell carcinoma) and 23 in the control group.
  Interventions: Procedure: Tumor removal
- Control group: 55 patients were included in the study : 32 in the cancer group (only squamous cell carcinoma) and 23 in the control group.
  Interventions: Procedure: Tumor removal

INTERVENTIONS:
Procedure: Tumor removal — Surgery

SUMMARY:
The main objective of our study was to determine the modifications of blood myostatin and activin A concentrations associated with head and neck cancers. Secondary objectives consisted in studying their influence on the occurrence of cachexia, bringing the proof of a tumoral secretion of these factors, and then determining the effect of tumor removal.

DETAILED DESCRIPTION:
Myostatin and activin A, two members of the superfamily TGF-β, have been shown to play a role on skeletal muscle mass regulation. In Humans, high plasma concentrations of activin A were observed in cancer patients, especially in cachectic subpopulations, suggesting their involvement in the development of cachexia.

55 patients were included in the study : 32 in the cancer group (only squamous cell carcinoma) and 23 in the control group. The patients underwent a complete nutritional assessment and multiple samples : blood before and 7 days after surgery, skeletal muscle biopsies, tumor biopsies. Plasma concentrations of myostatin, activin and follistatin were measured before and after tumor removal surgery. Concentrations of myostatin, activin and follistatin were also measured in an incubation medium of a tumor biopsy. Activin A and follistatin plasma concentrations were significantly increased in the cancer group (320 vs. 203 pg/ml ; p <0.001) (3593 vs 2148 pg/ml ; p <0.001), while myostatin plasma concentration was significantly decreased in this group (1542 vs. 2100 pg/ml ; p = 0.010). Surprisingly, data of the 7th postoperative day showed an increase in plasma activin A concentration (379 vs 320 pg /ml ; p <0.001) while concentrations of myostatin and follistatin were not modified. A high postoperative systemic inflammation is one hypothesis to explain these later results. Myostatin, activin A and follistatin proteins were systematically detected in the medium of tumor a 48 hour-incubation period, providing a strong proof of the tumor production of these factors by squamous cell carcinoma. The activin A/myostatin/follistatin is modified in the context of head and neck cancer. Activin A particularly seems to play a role in the occurrence of cachexia while follistatin could have a protective role for skeletal muscle mass. This system could aimed in therapeutic ways to reduce cachexia in a context of cancer in order to improve the quality of life and survival of patients.

ELIGIBILITY:
Inclusion Criteria:

For case group :

* head and neck cancer
* squamous cell carinoma only
* head and neck surgery chosen as treatment of cancer
* age 18-75

For control group :

* Neck surgery for non oncologic disease
* age 18-75

Exclusion Criteria:

* heart failure, respiratory failure (requiring a long-term oxygen therapy), chronic renal failure (MDRD clearance < 60 ml/min), moderate or severe chronic obstructive pulmonary disease and insulin-dependent diabeta for the two groups
* cachexia for control group

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 55 patients were included in the study : 32 in the cancer group (only squamous cell carcinoma) and 23 in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Measure of plasma activin A (pg/ml) | at day 1
  determine the modifications of blood myostatin and activin A concentrations associated with head and neck cancers
Measure of plasma follistation (pg/ml) | at day 1
  determine the modifications of blood myostatin and activin A concentrations associated with head and neck cancers
Measure of plasma myostatin (pg/ml) | at day 1
  determine the modifications of blood myostatin and activin A concentrations associated with head and neck cancers

SECONDARY OUTCOMES:
Influence on the occurrence of cachexia | at day 1
  Bringing the proof of a tumoral secretion of these factors, and then determining the effect of tumor removal.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne, France